CLINICAL TRIAL: NCT00124839
Title: Evaluation of the Efficacy of the Opioid Antagonist Naltrexone on the Incidence and Intensity of Flashbacks and Dissociative States in Patients With Borderline Personality Disorder
Brief Title: Naltrexone in Borderline Personality Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties in recruiting enough subjects
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Naltrexon-BPS
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Borderline Personality Disorder
Keywords: Dissociation; Flashbacks; Self-injurious behavior
MeSH Terms: conditions — Borderline Personality Disorder; Dissociative Disorders; Self-Injurious Behavior | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Other): Blinded sequential administration: naltrexon 50 mg (3 weeks)- placebo (3 weeks)- placebo (1 week)
  Interventions: Drug: Naltrexone
- 2 (Other): Blinded sequential administration: 200mg naltrexone (3 weeks) - placebo (3 weeks)- placebo (1 week)
  Interventions: Drug: Naltrexone
- 3 (Other): Blinded sequential administration: placebo (3 weeks) - 200mg naltrexone (3 weeks) - placebo (1 week)
  Interventions: Drug: Naltrexone
- 4 (Other): Blinded sequential administration: placebo (3 weeks) - 50mg naltrexone (3 weeks) - placebo (1 week)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Daily oral administration (capsules): 50mg naltrexone and placebo or 200mg naltrexone and placebo or placebo and naltrexon 50mg or placebo and 200mg naltrexone

SUMMARY:
The purpose of this study is to investigate whether naltrexone reduces the intensity and duration of flashbacks and dissociative states in patients with borderline personality disorder.

ELIGIBILITY:
Inclusion Criteria:

* In- and Outpatients:Borderline personality disorder according to the Diagnostic and Statistical Manual for Mental Disorders, 4.Edition (DSM IV)
* DES-(Dissociative Experience Scale)-score: > or equal 18 according to amendment4 (former value according to amendment 2 was > or equal 25).
* Urinary test of opiates negative
* No psychopharmacological treatment for two weeks prior to study (fluoxetine four weeks)
* No Lithium for two months

Exclusion Criteria:

* Lifetime diagnosis of psychotic disorder
* Current major depressive disorder (MDD)
* Lifetime diagnosis opioid dependence or current opioid abuse (10 to 7 days prior to study)
* Comedication with opioid analgetics
* Known naltrexone intolerance
* Liver disease
* Pregnancy and lactation period
* Other severe medical or neurological diseases
* Simultaneous participation in another study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Reduction of dissociative symptoms | End of 3rd week treatment of naltrexon

SECONDARY OUTCOMES:
Reduction of flashbacks | End of 3rd week treatment of naltrexone
Reduction of self-injurious behavior | End of 3rd week treatment of naltrexone
Reduction of psychopathology (depression, anxiety, anger, borderline symptoms) | End of 3rd week treatment of naltrexone
Safety regarding liver enzyme elevation | End of 3rd week treatment of naltrexone

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bohus, M.D., Study Director — University of Heidelberg, Central Institute of Mental Health Mannheim
Locations (5):
- Germany (5):
  - Dept. of Psychosomatic Medicine, Central Instiute of Mental Health, Mannheim, Baden-Würtemberg
  - Klinik Dr. Schlemmer GmbH, Center for Psychosomatic Medicine, Bad Wiessee, Bavaria
  - Inntalklinik Simbach am Inn, Simbach, Bavaria
  - Dept.of Psychiatry and Psychotherapy; Center of Neurology, Rostock, Mecklenburg-Vorpommern
  - Dept.of Psychiatry and Psychotherapy , Rheinische Kliniken Köln, Cologne, North Rhine-Westphalia

REFERENCES:
- [Background] Schmahl C, Bohus M. [Treatment of dissociative symptoms in borderline personality disorder with naltrexone: supplementary comments]. Nervenarzt. 2000 May;71(5):427. doi: 10.1007/s001150050582. No abstract available. German. PMID 10846724
- [Background] Bohus MJ, Landwehrmeyer GB, Stiglmayr CE, Limberger MF, Bohme R, Schmahl CG. Naltrexone in the treatment of dissociative symptoms in patients with borderline personality disorder: an open-label trial. J Clin Psychiatry. 1999 Sep;60(9):598-603. doi: 10.4088/jcp.v60n0906. PMID 10520978
- [Background] Schmahl C, Stiglmayr C, Bohme R, Bohus M. [Treatment of dissociative symptoms in borderline patients with naltrexone]. Nervenarzt. 1999 Mar;70(3):262-4. doi: 10.1007/s001150050431. German. PMID 10231814
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174